CLINICAL TRIAL: NCT05217576
Title: NBM-200 Clinical Study in Blood Donation Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OneBlood, Inc. (Other)
Collaborators: OrSense, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OrSense-001
Record Dates: First submitted 2021-09-09; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Hemoglobin H

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Comparison (Other): Comparison study:
  The participants (at least 300) will be tested once with each of the 3 devices. First, a measurement with the NBM-200 will be performed according to the user manual. The best finger to use, in order of preference: 1) right thumb 2) left thumb 3) right index 4) left index.
  The POC capillary test will follow the NBM-200 test, and the venous test will be performed last. A venous blood sample will be obtained from all participants in the comparison study, even if a subject is designated to donate and is deferred from donation because of low hemoglobin.
  Interventions: Device: NBM-200
- Precision A & B (Other): Precision study:
  1. At least 12 subjects will be tested 6 consecutive times with the NBM-200, on either the right or left thumb, and then 6 times with the capillary device (with a separate finger-prick for each test).
  2. At least 3 males and 3 females at 2 study sites (total of 12), preferably with hemoglobin levels close to the cutoff levels of 12.5 g/dL for females and 13 g/dL for males. Each subject will be tested on each of their right and left thumbs and indices (4 fingers) using at least two operators and two NBM-200 instruments on each finger.
  A laboratory test with venous blood is not required for participants in the precision study.
  Interventions: Device: NBM-200

INTERVENTIONS:
Device: NBM-200 — Finger Prick and Venipuncture
  Other Names: HemoCue-301-Hb

SUMMARY:
The NBM-200 is a portable Hemoglobin and oximetry monitor, based on occlusion spectroscopy technology, for non-invasive spot checking of hemoglobin (Hb), estimated Hematocrit (Hct), SpO2 and pulse rate.

The NBM-200 includes a reusable ring-shaped sensor probe that fits on the patient's finger, and a portable desktop monitor that calculates and displays the measurement result.

The sensor probe consists of a multi-wavelength optical measuring system and inflatable cuff employing pneumatic tissue manipulation. Blood flow in the finger can be briefly occluded and the resulting changes in its optical behavior are analyzed to provide accurate measurements of Hb.

DETAILED DESCRIPTION:
The proposed study plan will support a 510(k) submission for the non-invasive NBM-200 system with a blood bank indication. In accordance with the agency's suggestion, OrSense plans to use as a predicate an FDA-cleared blood analyzer with a hemoglobin test method that is traceable to the cyanmethemoglobin method or that was standardized and calibrated using the International Council for Standardization in Hematology (ICSH) hemoglobin standard, e.g., the HemoCue-301 or EKF's Hemo Control Hemoglobin Measurement System. OrSense further plans to use the cleared NBM-200 (K142209) as a reference device. Clinical data will be collected in a blood donor population using 3 methods to check hemoglobin (Hb): (1) the non-invasive NBM-200 system; (2) a point-of-care device based on finger sticks that is FDA-cleared for use in blood banks, such as the HemoCue or EKF device; and (3) a laboratory analyzer based on venous blood samples.

Participants will be recruited via email and during their visit to the designated donor rooms.

ELIGIBILITY:
Inclusion Criteria:

* Regular donors and volunteers

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Bias | 24 hours
  The mean bias between the NBM-200 and HemoCue readings and the laboratory reference

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Palm Harbor Donor Center, Palm Harbor, Florida
  - OneBlood St. Pete Main Donor Center, St. Petersburg, Florida
  - Tampa- Dale Mabry OneBlood Donor Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
At the conclusion of the study, the data will be published in reputable clinical journals.